CLINICAL TRIAL: NCT00800254
Title: Early Neuromuscular Electrical Stimulation For Quadriceps Muscle Activation Deficits Following Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American College of Rheumatology Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0074; K23AG029978-01A2 (NIH)
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis
Keywords: electrical stimulation; total knee arthroplasty; quadriceps; muscle; arthroscopy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular Electrical Stimulation (NMES) (Experimental)
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- Standard Rehabilitation Protocol (Active Comparator)
  Interventions: Other: Standard Rehabilitation Protocol

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — NMES 20 minutes twice a day for 6 weeks plus standard physical therapy
  Arms: Neuromuscular Electrical Stimulation (NMES)
Other: Standard Rehabilitation Protocol — Standard physical therapy for 8 weeks after surgery
  Arms: Standard Rehabilitation Protocol

SUMMARY:
The purpose of this study is to determine whether early intervention with neuromuscular electrical stimulation (NMES) for muscle strengthening immediately after total knee arthroplasty (TKA) is more effective than voluntary exercise alone in countering changes in quadriceps muscle activation, force production, and function in older adults.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic degenerative joint disease that disables about 10% of people over the age of 60 and compromises the quality of life of more than 20 million Americans. To alleviate pain and disability associated with knee OA, over 400,000 total knee arthroplasty (TKA) are performed each year in the United States, and future projections indicate that by the year 2030, more than 750,000 TKAs will be performed per year. While TKA reliably reduces pain and improves function, the recovery of force and function to normal levels is rare, which predisposes patients to future disability with increasing age. A month after TKA, impairments in quadriceps force are predominantly due to reflex inhibition, but are also influenced, to a lesser degree, by muscle atrophy. Neuromuscular electrical stimulation (NMES) may offer a promising alternative approach to override quadriceps reflex inhibition and prevent muscle atrophy to restore normal quadriceps muscle function more effectively than voluntary exercise alone, especially when applied within the first days after surgery.

The overall goal of this study is to evaluate the efficacy of NMES initiated 48hrs after TKA as an adjunct to standard rehabilitation. NMES is expected to more effectively restore normal quadriceps muscle function to produce greater quadriceps force by decreasing reflex inhibition. Patients will be randomized into one of two rehabilitation groups: 1) the standard rehabilitation group or 2) standard rehabilitation + NMES.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years of age
* Scheduled for a primary unilateral TKA
* Cognitive status that allows patients to consistently comprehend and repeat back directions regarding the details of the study

Exclusion Criteria:

* History of uncontrolled hypertension or uncontrolled diabetes
* Body mass index greater than 35 kg/m^2
* Neurological, vascular or cardiac problems that significantly limit function
* Moderate or severe osteoarthritis or other orthopedic conditions in the non-operated lower extremity that limit function

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens, MPT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCD Physical Therapy Program, Aurora, Colorado, United States

REFERENCES:
- [Background] Mintken PE, Carpenter KJ, Eckhoff D, Kohrt WM, Stevens JE. Early neuromuscular electrical stimulation to optimize quadriceps muscle function following total knee arthroplasty: a case report. J Orthop Sports Phys Ther. 2007 Jul;37(7):364-71. doi: 10.2519/jospt.2007.2541. PMID 17710905
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Derived] Stevens-Lapsley JE, Balter JE, Wolfe P, Eckhoff DG, Schwartz RS, Schenkman M, Kohrt WM. Relationship between intensity of quadriceps muscle neuromuscular electrical stimulation and strength recovery after total knee arthroplasty. Phys Ther. 2012 Sep;92(9):1187-96. doi: 10.2522/ptj.20110479. Epub 2012 May 31. PMID 22652985
- [Derived] Stevens-Lapsley JE, Balter JE, Wolfe P, Eckhoff DG, Kohrt WM. Early neuromuscular electrical stimulation to improve quadriceps muscle strength after total knee arthroplasty: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):210-26. doi: 10.2522/ptj.20110124. Epub 2011 Nov 17. PMID 22095207

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Rehabilitation Protocol (Control): Standard Rehabilitation Protocol: Standard physical therapy for 8 weeks after surgery
Period: Overall Study
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Started | 35 | 31
3.5 Weeks Post-operatively | 31 | 31
Completed | 30 | 25
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control) | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.1) | 64.8 (7.7) | 65.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 15 | 15 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.9) | 31.2 (4.2) | 29.2 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Isometric Quadriceps Muscle Torque 3.5 Weeks Post-operatively
Description: A HUMAC NORM electromechanical dynamometer was used to measure isometric torque generation in quadriceps muscle stabilized with 60 degrees of knee flexion.
Time Frame: Baseline through 3.5 weeks
Population: The Participant Flow represents overall study enrollment and withdrawals. In some cases, patients may have returned for testing, but been unable to complete every test due to time constraints, fatigue, or in some cases, inability.
Measure: Mean (Standard Error); unit: change in N-m/kg
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 35 | 31
change in N-m/kg | -0.40 (0.05) | -0.67 (0.06)
Statistical Analysis 1: Comparison: Neuromuscular Electrical Stimulation (NMES) vs Standard Rehabilitation Protocol (Control); Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in Isometric Quadriceps Muscle Torque 1-Year Post-operatively
Description: as for outcome 1
Time Frame: Baseline through 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in N-m/kg
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 30 | 25
change in N-m/kg | 0.33 (0.52) | 0.18 (0.43)

3. Secondary Outcome: Functional Performance Measure: Six-Minute Walk Test [6MWT]) at 3.5 Weeks Post-operatively
Description: The 6MWT assesses the total distance in meters a patient walks at a self-selected pace over a 6 minute interval.
Time Frame: 3.5 weeks post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 31 | 24
meters | 390.1 (92.4) | 295.3 (103.4)
Statistical Analysis 1: Comparison: Neuromuscular Electrical Stimulation (NMES) vs Standard Rehabilitation Protocol (Control); Test type: Superiority or Other; p < 0.003, ANCOVA

4. Secondary Outcome: Functional Performance Measure: Timed "Up & Go" Test [TUG] at 3.5 Weeks Post-operatively
Description: The TUG assesses time in seconds to rise from an armchair, walk 3 meters, turn around, and return to sitting in the same chair without physical assistance.
Time Frame: 3.5 weeks post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 31 | 28
seconds | 10.4 (3.8) | 13.9 (4.5)

5. Secondary Outcome: Functional Performance Measure: Stair-Climbing Test [SCT] at 3.5 Weeks Post-operatively
Description: The SCT assesses the time it takes for a patient to ascend a flight of stairs, turn around, and descend the same flight of stairs.
Time Frame: 3.5 weeks post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 30 | 28
seconds | 25.2 (10.4) | 39.3 (13.9)

6. Secondary Outcome: Functional Performance Measure: Six-Minute Walk Test [6MWT]) at 1 Year Post-operatively
Description: The 6MWT assesses the total distance in meters a patient walks at a self-selected pace over a 6 minute interval.
Time Frame: 1 year post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 29 | 25
meters | 524.6 (81.6) | 477.8 (94.0)

7. Secondary Outcome: Functional Performance Measure: Timed "Up & Go" Test [TUG] at 1 Year Post-operatively
Description: as for outcome 4
Time Frame: 1 year post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 29 | 25
seconds | 6.7 (1.7) | 8.3 (2.8)

8. Secondary Outcome: Functional Performance Measure: Stair-Climbing Test [SCT] at 1 Year Post-operatively
Description: as for outcome 5
Time Frame: 1 year post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol (Control)
Number analyzed (Participants) | 29 | 25
seconds | 11.5 (4.3) | 14.8 (9.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of 1 year.
Arm/Group | Neuromuscular Electrical Stimulation (NMES) | Standard Rehabilitation Protocol
Serious Adverse Events (participants affected / at risk) | 3/35 | 3/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neuromuscular Electrical Stimulation (NMES) (N=35) | Standard Rehabilitation Protocol (N=31)
Post-op complication (Surgical and medical procedures) | 1 | 0
DVT (Blood and lymphatic system disorders) | 1 | 0
Severe Sciatica (Nervous system disorders) | 1 | 0
Infection in the knee (Infections and infestations) | 0 | 1
C-Diff infection (Infections and infestations) | 0 | 1
TKA revision (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes